CLINICAL TRIAL: NCT01619163
Title: Phase 4 Study of Low Dose Prednisolone for Knee Osteoarthritis
Brief Title: Prednisolone for Pain Reduction in Knee OA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, Professor of Rheumatology, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: alexmed11662452
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: Prednisolone,; pain,; inflammation,; mobility; Function
MeSH Terms: conditions — Pain; Inflammation | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisolone (Experimental)
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Prednisolone — low dose, 7.5 mg/day
  Arms: prednisolone

SUMMARY:
Background: Osteoarthritis (OA), a common disabling condition, is the commonest type of arthritis worldwide. Knee OA is the 4th leading cause of disability in women. Pain is the leading symptom and is often chronic in nature leading to significant morbidity and decreased quality of life. Synovitis is prevalent in knee OA and treatment to relieve this synovitis may reduce pain.

Objectives: A randomized double-blind placebo-controlled trial will be conducted to assess whether 6 weeks of daily low dose oral prednisolone will improve pain, mobility and systemic low-grade inflammation, in the short term and to determine if it sustained long term at 12 weeks in older adults with moderate to severe knee OA.

Methods: 125 community-dwelling older adults aged 65 years and above with primary knee OA diagnosed according to the ACR criteria for diagnosis of primary OA of the knee will berandomized 1:1. Sixty three will receive 7.5 mg/day of prednisolone and 62 will receive placebo together with their usual therapy for 6 weeks. The primary outcome measure will be pain reduction. Secondary outcome measures will be reduction in systemic inflammation and improvements in physical functioning scores. Alterations in dosage of analgesic/NSAID drugs used will be recorded. Safety and tolerability were also assessed. Data will be collected at baseline, 6 weeks and at 12 weeks to determine any change in results from those obtained at 6 weeks. Exclusion criteria will include any inflammatory or serious medical condition.

Knee OA will be documented by radiographic examination using the Kellgren-Lawrence scale. Symptomatic OA will be defined as the need to take NSAIDs daily and LequesneAlgofunctional Index (LFI)score > 4. Clinical assessment will be include: Visual Analogue Pain Scale (VAS, 0-100), self-reported physical function as measured with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), WOMAC pain and stiffness scores, and six-minute walk distance (6MWD). All patients will undergo a physical examination and will be questioned about the number of flares, pain and analgesic use. Blood samples will be collected and serum levels of IL-1, IL-6, TNF-alpha and hsCRP will be measured in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 65 years and above with primary knee OA diagnosed according to the ACR criteria for diagnosis of primary OA of the knee

Exclusion Criteria:

* Any inflammatory or serious medical condition

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 6 weeks
  The primary outcome measure was pain reduction.

SECONDARY OUTCOMES:
Reduction in systemic inflammation and improvements in physical functioning scores. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt

REFERENCES:
- [Derived] Abou-Raya A, Abou-Raya S, Khadrawi T, Helmii M. Effect of low-dose oral prednisolone on symptoms and systemic inflammation in older adults with moderate to severe knee osteoarthritis: a randomized placebo-controlled trial. J Rheumatol. 2014 Jan;41(1):53-9. doi: 10.3899/jrheum.130199. Epub 2013 Dec 1. PMID 24293578 (Retraction: PMID 30504483 J Rheumatol. 2018 Dec;45(12):1713)